CLINICAL TRIAL: NCT00260572
Title: Outcomes After Medical and Surgical Treatment of Gastroesophageal Reflux Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, James Luketich, MD, University of Pittsburgh
Other Study IDs: STUDY20050057
Record Dates: First submitted 2005-11-28; First posted 2005-12-01 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-02

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; nissen; fundoplication; reflux; toupet; QOL; dyspepsia; heartburn; Patients with reflux symptoms for at least 6 months; Patients scheduled for lap nissen or toupet fundoplication; Reflux diagnosed by either endoscopy, upper GI, or 24hr. pH (numeric scale used to specify the acidity of gastric contents); On or starting treatment with PPI or pro-motility agents
MeSH Terms: conditions — Gastroesophageal Reflux; Dyspepsia; Heartburn | interventions — Quality of Life; Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Questionnaires to evaluate QOL — Questionnaire to evaluate QOL administered preoperatively and postoperatively at set intervals.
Behavioral: Questionnaires to evaluate heartburn and quality of life — Questionnaires to evaluate heartburn and quality of life administered preoperatively and at set intervals postoperatively.
Behavioral: Questionnaire to evaluate satisfaction with treatment — Questionnaire administered postoperatively at set intervals.
Behavioral: Questionnaire to evaluate presence or absence of pain — Questionnaire administered preoperatively and at set intervals postoperatively.

SUMMARY:
The aims of this study are to create a prospective data base to evaluate the long term outcomes of medical and surgical treatment of gastroesophageal reflux disease (GERD); to measure standard outcomes as well as patient derived outcomes such as general and disease specific quality of life (QOL) issues and patient satisfaction; to refine the parameters that may identify patients who will benefit from surgery for GERD; and to identify possible determinants of failure of both medical and surgical treatments of reflux.

DETAILED DESCRIPTION:
GERD is a significant public health problem and when it is severe it may have a considerable impact on patients' QOL. Relatively new treatments such as proton pump inhibitors (PPI) and laparoscopic fundoplication (wrapping or gathering the stomach around the lower end of the esophagus to reduce or prevent reflux) are now available. Patient derived outcomes such as QOL and satisfaction are rarely taken into consideration when evaluating such new treatments. Outcome analysis of the results of medical and surgical treatments using an ongoing database of patients will enhance our ability to treat patients with GERD.

This study's goal is to build a database to collect the outcome information on patients who are having medical or surgical treatment of GERD. In addition we want to measure standard outcomes such as morbidity, mortality, medication use and patient derived outcomes such as general and disease specific QOL, and patient satisfaction with the treatment. We also want to assess if and how long QOL is improved by medical and surgical treatment methods. In addition we want to see if low QOL scores on medical treatment as well as the standard medical criteria can help to identify which patients may benefit from surgical (an operation) rather than the medical treatment. It is hoped that we can also identify which factors might predict or help to determine which patients will have failure of both medical and surgical treatments of GERD. Using this information we want to identify if a psychological profile done before treatment will influence or predict the outcomes of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with reflux symptoms present for at least 6 months, caused by documented reflux. Reflux symptoms include:

  * heartburn
  * acid regurgitation
  * waterbrash
  * non-cardiac chest pain
  * dyspepsia
* Reflux diagnosis either by endoscopy, upper gastrointestinal (GI), or 24 hour pH.
* Patients scheduled for surgical management of GERD and/or hiatal hernia
* Patients currently or commencing treatment with at least proton pump inhibitors or pro-motility agents.

Exclusion Criteria:

* Patients unable to comprehend or complete the QOL instruments.
* Patients less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of reflux seeking treatment in a physician's office.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 1999-04; Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Luketich, MD, Principal Investigator — Department of Cardiothoracic Surgery
Locations (1):
- UPMC Department of Cardiothoracic Surgery, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided